CLINICAL TRIAL: NCT03912467
Title: Prevalence of Pressure Ulcers Among Critically Ill Patients and Factors Associated With Their Occurrence in the ICU
Acronym: PRESSURE
Status: Completed | Type: Observational
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: PRESSURE
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Pressure Ulcer; Critical Care; Intensive Care Unit Syndrome
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pressure Ulcer Evaluation — Patient was evaluated according to presence of pressur ulcer or not

SUMMARY:
The prevalence of and risk factors for pressure ulcers (PUs) in critically ill patients have been poorly studied. The main objective of this study was to describe the prevalence of PUs in critically ill patients. Secondary objectives were to describe PUs, means of prevention of PUs, and factors associated with occurrence of PUs in the ICU.

DETAILED DESCRIPTION:
Pressure ulcers (PUs) among hospitalized patients are associated with a poor prognosis and with a high cost of care. Hospitalization in the ICU is a context where there is a high risk of occurrence of PUs, prevention of which is a priority for ICU teams caring for critically ill patients. However, the literature is inconclusive regarding the prevalence of PUs among critically ill patients and the associated risk factors. The main objective of this study was to describe the prevalence of PUs among critically ill patients hospitalized in the ICU. Secondary objectives were to describe means of prevention of PUs in the ICU and the characteristics of PUs, and to identify factors either related to the ICU or patient characteristics associated with occurrence of PUs in the ICU.

ELIGIBILITY:
The inclusion criteria were :

* hospitalization in the ICU
* age ≥ 18 years.

The exclusion criterion was:

- refusal to participate in the study by the patient or by the patient's family when the patient was unable to consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient in Critical Care during study day.
Sampling Method: Non-Probability Sample
Enrollment: 1228 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Pressure Ulcer Presence on the study day | Through study completion, an average of 1 day
  Presence (1) or absence (0) of pressure ulcer (however grade of pressure ulcer) during the study period which is a 1 Day Study Prevalence

SECONDARY OUTCOMES:
Grade of Pressure Ulcer on the study day | Through study completion, an average of 1 day
  Grade (from 1 to 4) of pressure ulcer during the study period which is a 1 Day Study Prevalence
Area of Pressure Ulcer on the study day | Through study completion, an average of 1 day
  Area on the patient's body of pressure ulcer during the study period which is a 1 Day Study Prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Gael Piton, MD, PhD, Study Chair — French Intensive Care Society
Locations (60):
- France (60):
  - Hôpital Saint-Esprit, Agen
  - CHU d'Angers, Angers
  - Hopital Privé d'Antony, Antony
  - Hopital Mercy, Ars-Laquenexy
  - Hopital Nord Franche Comté, Belfort
  - Hopital Avicenne, Bobigny
  - CHU Pellegrin, Bordeaux
  - Hopital St-Andre, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - HIA Clermont Tonnerre, Brest
  - Hopital Antoine Beclere, Clamart
  - HIA Percy, Clamart
  - Hopital Louis Mourier, Colombes
  - Groupe Hospitalier Sud Ile de France, Corbeil-Essonnes
  - Clinique des Cèdres, Cornebarrieu
  - CHU Henri Mondor, Créteil
  - CHU Dijon Bourgogne, Dijon
  - Hopital Simone Veil, Eaubonne
  - Hopital Raymond Poincare, Garches
  - CHU Grenoble Alpes, Grenoble
  - Grand Hopital de l'Est Francilien, Jossigny
  - CHU Réunion Saint Pierre, La Réunion
  - CHU Kremlin-Bicetre, Le Kremlin-Bicêtre
  - Hopital Roger Salengro, Lille
  - HIA Desgenettes Lyon, Lyon
  - Groupe Hospitalier Edouard Herriot, Lyon
  - Hopital Francois Quesnay, Mantes-la-Jolie
  - Hopital Européen Marseille, Marseille
  - CHU Marseille Hopital Nord, Marseille
  - Hopital de la Timone, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - GHIRM, Montfermeil
  - CHU Lapeyronie, Montpellier
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hopital Laennec, Nantes
  - Hopital l'Archet, Nice
  - CHU Nimes, Nîmes
  - Hopital St Louis, Paris
  - GH Diaconnesses Croix Saint Simon, Paris
  - La Pitié Salpetriere, Paris
  - Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Necker Enfants Malades, Paris
  - CHU Robert Debré, Paris
  - HEGP, Paris
  - Hopital Tenon, Paris
  - CHU Poitiers, Poitiers
  - Hopital Privé Claude Galien, Quincy-sous-Sénart
  - Hopital Delafontaine, Saint-Denis
  - Clinique de l'Union, Saint-Jean
  - HIA Béjin, Saint-Mandé
  - Hopital Saint Clair, Sète
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - Hopital Privé du Vert Galan, Tremblay-en-France
  - Hopital Jean Bernard, Valenciennes
  - Institut Gustave Roussy, Villejuif
  - HIA Robert Pique, Villenave-d'Ornon
  - Hopital Privé du Val d'Yerres, Yerres

IPD SHARING:
Plan to Share IPD: No